CLINICAL TRIAL: NCT04022239
Title: Post-Transplant Bendamustine (PT-BEN) for GVHD Prophylaxis
Brief Title: Bendamustine With or Without Cyclophosphamide in Preventing GVHD in Patients Undergoing Stem Cell Transplant
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0972; NCI-2019-03900 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0972 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm
MeSH Terms: interventions — Stem Cell Transplantation; Bendamustine Hydrochloride; Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine; Melphalan; Mycophenolic Acid; Rituximab; CT-P10; Tacrolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Schedule I (non-lymphoma) (Experimental): Patients receive fludarabine IV over 1 hour on days -5 to -2, melphalan IV over 30 minutes on days -5 and -4, and undergo TBI on day -1 and stem cell transplantation IV over 2-6 hours on day 0. Depending on when the trial was joined, patients receive cyclophosphamide IV over 3 hours or bendamustine IV over 30-60 minutes or cyclophosphamide IV over 3 hours and bendamustine IV over 30-60 minutes on day 3. Patients also receive bendamustine IV over 30-60 minutes on day 4. Beginning day 5, patients receive tacrolimus IV followed by PO QD or BID for 6 months and mycophenolate mofetil PO TID until day 100. Beginning day 7, patients receive filgrastim-sndz SC QD until blood cell levels return to normal.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Bendamustine; Drug: Cyclophosphamide; Biological: Filgrastim-sndz; Drug: Fludarabine; Drug: Melphalan; Drug: Mycophenolate Mofetil; Drug: Tacrolimus; Radiation: Total-Body Irradiation
- Schedule II (lymphoid malignancies) (Experimental): Patients receive fludarabine IV over 1 hour, bendamustine IV over 30-60 minutes on days -5 to -3 and undergo TBI on day -1 and stem cell transplantation over 2-6 hours on day 0. Depending on when the trial was joined, patients receive cyclophosphamide IV over 3 hours or bendamustine IV over 30-60 minutes or cyclophosphamide IV over 3 hours and bendamustine IV over 30-60 minutes on day 3. Patients also receive bendamustine IV over 30-60 minutes on day 4. Beginning day 5, patients receive tacrolimus IV followed by PO QD or BID for 6 months and mycophenolate mofetil PO TID until day 100. Beginning day 7, patients receive filgrastim-sndz SC QD until blood cell levels return to normal. CD20+ patients receive rituximab IV over 4-6 hours on days -13, -6, 1, and 8.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Bendamustine; Drug: Cyclophosphamide; Biological: Filgrastim-sndz; Drug: Fludarabine; Drug: Mycophenolate Mofetil; Biological: Rituximab; Drug: Tacrolimus; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo stem cell transplantation
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Drug: Bendamustine — Given IV
  Other Names: SDX-105
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Biological: Filgrastim-sndz — Given SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Zarxio
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
  Arms: Schedule I (non-lymphoma)
Drug: Mycophenolate Mofetil — Given PO
  Other Names: CellCept; MMF
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
  Arms: Schedule II (lymphoid malignancies)
Drug: Tacrolimus — Given IV and PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: SCT_TBI; TBI; Total Body Irradiation; Whole Body Irradiation; Whole-Body Irradiation

SUMMARY:
This phase I/II trial studies the side effects and best dose of bendamustine when given with or without cyclophosphamide in preventing graft versus host disease (GVHD) in patients undergoing stem cell transplant. Drugs used in chemotherapy, such as bendamustine and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy and total body irradiation before or after a stem cell transplant helps kills cancer cells that are in the body and helps make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow. Sometimes, the transplanted cells from a donor can attack the body's normal cells called GVHD. Giving tacrolimus, mycophenolate mofetil, and filgrastim after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the safety of substituting the standard post-transplant cyclophosphamide (PT-CY) given on day +3 and +4 with post-transplant bendamustine (PT-BEN) in patients undergoing HLA-mismatched hematopoietic cell transplantation.

SECONDARY OBJECTIVES:

I. To evaluate treatment-related mortality. II. To assess acute and chronic graft-versus-host disease (GVHD). III. To assess overall survival, progression-free survival and relapse rates. IV. To evaluate the risk of acute cystitis. V. To evaluate immune reconstitution after transplantation.

OUTLINE: This is a dose-escalation study of bendamustine. Patients are assigned to 1 of 2 treatment schedules.

SCHEDULE I (NON-LYMPHOMA): Patients receive fludarabine intravenously (IV) over 1 hour on days -5 to -2, melphalan IV over 30 minutes on days -5 and -4, and undergo total body irradiation (TBI) on day -1 and stem cell transplantation IV over 2-6 hours on day 0. Depending on when the trial was joined, patients receive cyclophosphamide IV over 3 hours or bendamustine IV over 30-60 minutes or cyclophosphamide IV over 3 hours and bendamustine IV over 30-60 minutes on day 3. Patients also receive bendamustine IV over 30-60 minutes on day 4. Beginning day 5, patients receive tacrolimus IV followed by orally (PO) once daily (QD) or twice daily (BID) for 6 months and mycophenolate mofetil PO thrice daily (TID) until day 100. Beginning day 7, patients receive filgrastim-sndz subcutaneously (SC) QD until blood cell levels return to normal.

SCHEDULE II (LYMPHOID MALIGNANCIES): Patients receive fludarabine IV over 1 hour, bendamustine IV over 30-60 minutes on days -5 to -3 and undergo TBI on day -1 and stem cell transplantation over 2-6 hours on day 0. Depending on when the trial was joined, patients receive cyclophosphamide IV over 3 hours or bendamustine IV over 30-60 minutes or cyclophosphamide IV over 3 hours and bendamustine IV over 30-60 minutes on day 3. Patients also receive bendamustine IV over 30-60 minutes on day 4. Beginning day 5, patients receive tacrolimus IV followed by PO QD or BID for 6 months and mycophenolate mofetil PO TID until day 100. Beginning day 7, patients receive filgrastim-sndz SC QD until blood cell levels return to normal. CD20+ patients receive rituximab IV over 4-6 hours on days -13, -6, 1, and 8.

After completion of study treatment, patients are followed weekly for 3 months, every 3 months in year 1, and every 6 months in year 2.

ELIGIBILITY:
Inclusion Criteria:

* Patient with hematologic malignancies.
* Donor: Matched sibling, matched unrelated, mismatched or haploidentical
* Zubrod performance 0 to 2 or Karnofsky of at least 60.
* Adequate organ function at time of study entry:

  1. Creatinine less than or equal to 1.6 mg/dL and creatinine clearance >/= 30 ml/min. Creatinine clearance will be calculated using the Cockcroft-Gault equation
  2. Total bilirubin less than < 1.5 x UNL
  3. SGPT < 2.5 x ULN
  4. Ejection fraction >/= 40%
  5. FEV1, FVC and DLCO >/= 40%
* Female patients of childbearing potential must agree to use an effective method of birth control while on study and for 6 months after the last dose of bendamustine. Male patients with female partners of childbearing potential must agree to use an effective method of birth control while on study and for 3 months after the last dose of bendamustine.

Exclusion Criteria:

* Pregnant or nursing women.
* Known to be HIV positive
* Active and uncontrolled disease/infection
* Unable or unwilling to sign consent
* Current active hepatic or biliary disease (with exception of Gilbert's syndrome)
* Active hepatitis B or C.
* Toxicities (grade > 1) unresolved from prior treatment (including chemotherapy, targeted therapy, immunotherapy, experimental agents radiation, or surgery.
* Patients with standard risk acute leukemia in first complete remission and patients with chronic myeloid leukemia in first chronic will be excluded during escalated phase.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose level (MTDL) (Phase I) | Up to 30 days
  Will employ the time-to-event Bayesian optimal interval design to find the MTDL. After the trial is completed, the MTDL will be selected based on isotonic regression as specified in Yuan et al. Specifically, MTDL will be selected as the dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate. If there are ties, the higher dose level when the isotonic estimate is lower than the target toxicity rate will be selected and the lower dose level when the isotonic estimate is greater than or equal to the target toxicity rate will be selected.
Dose-limiting toxicity (Phase I) | Up to 100 days
Incidence of adverse events (Phase II) | Up to 2 years
  The trial is continuously monitored for toxicity per the statistical design.

CONTACTS AND LOCATIONS:
Overall Officials: Issa F Khouri, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org